CLINICAL TRIAL: NCT02689076
Title: Regional Data Exchange to Improve Care for Veterans After Non-VA Hospitalization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 14-049
Record Dates: First submitted 2016-02-18; First posted 2016-02-23 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Patient Readmission; Adverse Drug Event; Cost
Keywords: Patient transfer; Patient care management; Health information exchange
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIE Notification plus Care Coordination (Experimental): VA provider notification of non-VA hospitalization via electronic health information exchange (HIE) plus post-hospital geriatric care transitions intervention
  Interventions: Other: HIE Notification; Other: Care transitions intervention
- HIE Notification alone (Active Comparator): VA provider notification of non-VA hospitalization via electronic health information exchange (HIE) followed by usual post-hospital care
  Interventions: Other: HIE Notification
- Usual Care (No HIE Notification and No Care Coordination) (No Intervention): Absence of VA provider notification of non-VA hospitalization via HIE plus Absence of post-hospital geriatric care transitions intervention [Usual Care]

INTERVENTIONS:
Other: HIE Notification — VA provider notification of non-VA hospitalization or ED visit via electronic health information exchange
  Arms: HIE Notification alone; HIE Notification plus Care Coordination
Other: Care transitions intervention — Post-hospital geriatrics care transitions coordinator provides home visit and telephone support for 30 days after hospital discharge
  Arms: HIE Notification plus Care Coordination

SUMMARY:
Among older VA patients who have Medicare coverage, 43% use both VA and non-VA (Medicare-covered) services. VA and non-VA providers are often uninformed about encounters, treatments and test results provided in the other system. The overall objective of this project is to examine the impact of VA provider notification of non-VA hospitalization or emergency department (ED) visit using electronic health information exchange (HIE), along with provision of post-hospital care coordination services. The investigators will examine the impact of these approaches on preventing hospital readmission, increasing provider follow-up, improving patient's self-knowledge, and preventing medication errors. The investigators will also examine the effect of these approaches on VA and non-VA costs. Finally the investigators will examine the acceptance of these approaches among VA and non-VA providers. The study sample will consist of Veterans followed in geriatrics or primary care clinics at the Bronx and Indianapolis VAs who are older than 65. The investigators will monitor patients for non-VA hospital admission or ED visit using technology provided by health information exchange organizations. Patients will be assigned to enhanced or control treatment groups. For both groups the VA provider will receive an electronic notification of a non-VA hospital admission or ED visit if it occurs. For the enhanced group, a care transitions coordinator will deliver post-hospital coordination services during a home and/or VA facility visit and follow-up phone calls over 1 month. The investigators' analyses will compare effects of notification-plus-coordination versus notification-only on health care outcomes. The investigators will conduct interviews with intervention team members, patients, VA and non-VA staff, and other stakeholders to ascertain the barriers and facilitators to implementation of these approaches.

DETAILED DESCRIPTION:
Background: Among older VA patients who have Medicare coverage, 43% use both VA and non-VA (Medicare-covered) services. VA and non-VA providers are often uninformed about encounters, treatments and test results provided in the other system. In particular, the absent or delayed notification of a non-VA hospital encounter is a missed opportunity for the VA to provide post-hospital transitional care services that have been shown to be effective in preventing adverse events and hospital readmission after hospital discharge. Objectives: The overall objective of this project is to examine the effectiveness, cost, and implementation acceptance of VA provider notification of non-VA hospitalization or emergency department (ED) visit using electronic health information exchange (HIE), with or without provision of evidence-based post-hospital transitional care services. Specific Aim 1 is to examine the impact of these approaches on preventing hospital admission or readmission as the primary outcome, and, as secondary outcomes, increasing provider follow-up, improving patient's condition self-knowledge, and preventing medication errors after discharge. been shown to be effective in preventing adverse events and hospital readmission after hospital discharge.

Specific Aim 2 is to examine the effect of these approaches on VA and non-VA costs. Specific Aim 3 is to examine the acceptance of these approaches among VA and non-VA stakeholders.

Methods: The study sample consists of Veterans followed in geriatrics or primary care clinics at the Bronx and Indianapolis VAs who are older than 65. The investigators will monitor patients for non-VA hospital admission or ED visit using technology provided by regional HIE organizations (i.e., the Bronx Regional Health Information Organization and the Indiana Health Information Exchange). Patients will be cluster-randomized 1:1 to notification-plus-coordination or notification-only groups by PACT team, stratified by facility. For both groups the PACT provider will receive real-time notification of a non-VA hospital admission or ED visit if it occurs. For the notification-plus-coordination group, a care transitions coordinator will deliver coordination activities during a home and/or VA facility visit and via follow-up phone calls over 1 month. Coordination activities will consist of: reconciliation of and counseling on the patient's VA and non-VA medications, education on signs of condition worsening, coordination of VA and non-VA follow-up appointments, and counseling on communicating with VA and non-VA providers, using structured protocols. All information-gathering by the transitions coordinator will include the HIE as an information source. The notification-only group will receive usual care after the notification. Multivariable regression models will be estimated to compare effects of notification-plus-coordination versus notification-only on primary and secondary outcomes and costs (Aims 1 and 2). The investigators will conduct interviews with intervention team members, patients, VA and non-VA staff, and other stakeholders to ascertain the barriers and facilitators to implementation of these approaches (Aim 3).

ELIGIBILITY:
Inclusion Criteria:

* established patient in a Bronx VA or Indianapolis VA geriatrics or primary care clinic
* 65 years or older
* be consented in the local health information exchange
* have utilized any non-VA services in the previous two years, including:

  * nursing
  * lab
  * physician
  * pharmacy
  * and/or hospital services

Exclusion Criteria:

* Refusal to sign informed consent or consent to access local health information exchange
* Enrolled in hospice at baseline
* Enrolled in Geriatric Resources and Care for Elders (GRACE) program (Indianapolis) at baseline

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 796 (Actual)
Dates: Start 2016-03-14 (Actual); Primary Completion 2020-04-05 (Actual); Study Completion 2020-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth S Boockvar, MD MS, Principal Investigator — James J. Peters Veterans Affairs Medical Center
Locations (2):
- United States (2):
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana
  - James J. Peters VA Medical Center, Bronx, NY, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dixon BE, Boockvar KS. Event Notification in Support of Population Health: The Promise and Challenges from a Randomized Controlled Trial. Stud Health Technol Inform. 2017;245:1357. PMID 29295436
- [Result] Dixon BE, Schwartzkopf AL, Guerrero VM, May J, Koufacos NS, Bean AM, Penrod JD, Schubert CC, Boockvar KS. Regional data exchange to improve care for veterans after non-VA hospitalization: a randomized controlled trial. BMC Med Inform Decis Mak. 2019 Jul 4;19(1):125. doi: 10.1186/s12911-019-0849-1. PMID 31272427
- [Result] Franzosa E, Traylor MH, Aquino VG, Judon K, Schwartzkopf A, Dixon BE, Boockvar K. Care Team Members' Perceptions of an Informatics Intervention to Improve Geriatric Care Across Multiple sites. [Abstract]. Innovation in aging. 2020 Dec 16; 4(Supplement_1):519.
- [Result] Franzosa E, Traylor M, Judon KM, Guerrero Aquino V, Schwartzkopf AL, Boockvar KS, Dixon BE. Perceptions of event notification following discharge to improve geriatric care: qualitative interviews of care team members from a 2-site cluster randomized trial. J Am Med Inform Assoc. 2021 Jul 30;28(8):1728-1735. doi: 10.1093/jamia/ocab074. PMID 33997903
- [Result] Kartje R, Dixon BE, Schwartzkopf AL, Guerrero V, Judon KM, Yi JC, Boockvar K. Characteristics of Veterans With Non-VA Encounters Enrolled in a Trial of Standards-Based, Interoperable Event Notification and Care Coordination. J Am Board Fam Med. 2021 Mar-Apr;34(2):301-308. doi: 10.3122/jabfm.2021.02.200251. PMID 33832998
- [Result] Koufacos NS, May J, Judon KM, Franzosa E, Dixon BE, Schubert CC, Schwartzkopf AL, Guerrero VM, Traylor M, Boockvar KS. Improving Patient Activation among Older Veterans: Results from a Social Worker-Led Care Transitions Intervention. J Gerontol Soc Work. 2022 Jan;65(1):63-77. doi: 10.1080/01634372.2021.1932003. Epub 2021 May 30. PMID 34053407
- [Result] Dixon BE, Judon KM, Schwartzkopf AL, Guerrero VM, Koufacos NS, May J, Schubert CC, Boockvar KS. Impact of event notification services on timely follow-up and rehospitalization among primary care patients at two Veterans Affairs Medical Centers. J Am Med Inform Assoc. 2021 Nov 25;28(12):2593-2600. doi: 10.1093/jamia/ocab189. PMID 34597411
- [Result] Boockvar KS, Koufacos NS, May J, Schwartzkopf AL, Guerrero VM, Judon KM, Schubert CC, Franzosa E, Dixon BE. Effect of Health Information Exchange Plus a Care Transitions Intervention on Post-Hospital Outcomes Among VA Primary Care Patients: a Randomized Clinical Trial. J Gen Intern Med. 2022 Dec;37(16):4054-4061. doi: 10.1007/s11606-022-07397-5. Epub 2022 Feb 23. PMID 35199262

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone | Usual Care (No HIE Notification and No Care Coordination)
Started | 268 | 337 | 191
Completed | 87 | 115 | 191
Not Completed | 181 | 222 | 0
Not completed — Did not have a non-VA encounter during study period (includes death before a non-VA encounter) | 172 | 213 | 0
Not completed — Discharged from non-VA facility to long-term care facility for an indefinite period | 3 | 1 | 0
Not completed — Did not have an HIE match | 2 | 0 | 0
Not completed — Death during non-VA encounter | 2 | 5 | 0
Not completed — Provider declined to participate after participant assignment | 1 | 1 | 0
Not completed — Participant no longer active in VA system | 1 | 0 | 0
Not completed — Enrolled in GRACE or hospice during non-VA encounter | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone | Usual Care (No HIE Notification and No Care Coordination) | Total
Number analyzed (Participants) | 87 | 115 | 191 | 393
Age, Continuous [Mean (Standard Deviation); unit: Years] | 77.7 (8.5) | 76.3 (7.4) | 72.5 (7.1) | 74.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 8
  Male | 86 | 113 | 186 | 385
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 14 | 27 | 53
  Not Hispanic or Latino | 75 | 98 | 164 | 337
  Unknown or Not Reported | 0 | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Black or African American | 15 | 28 | 64 | 107
  White | 69 | 79 | 110 | 258
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 2 | 5 | 16 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 115 | 191 | 393
VA Hospital Utilization in Year Prior to Enrollment [Count of Participants; unit: Participants] | 9 | 16 | 33 | 58

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Hospital Readmission
Description: Percentage of patients with VA and non-VA hospital admission or readmission 90 days after non-VA hospital or ED discharge (or, if the patient is not discharged home, 90 days after discharge home from a rehabilitation facility)
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone | Usual Care (No HIE Notification and No Care Coordination)
Number analyzed (Participants) | 87 | 115 | 191
Participants | 23 | 21 | 35

2. Secondary Outcome: Number of Participants With Scheduled Follow-up
Description: VA follow-up visit with a VA provider (physician or nurse practitioner) within 30 days of non-VA hospital discharge or ED visit.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone | Usual Care (No HIE Notification and No Care Coordination)
Number analyzed (Participants) | 87 | 115 | 191
Participants | 35 | 37 | 39

3. Secondary Outcome: Number of High-risk Medication Discrepancies
Description: The number of discrepancies in medications classified as high risk for hospitalized older adults, including opioid analgesics, insulin, non-steroidal anti-inflammatory drugs, digoxin, antipsychotics, sedatives/hypnotics, and anticoagulants based on medical record review and patient or caregiver interview 30 days after non-VA hospital discharge.
Time Frame: 30 days
Population: Participants were included in the analysis who had a 30-day interview and answered the required questions. No participants in the Usual Care group are included in the analysis because they did not have a 30-day interview.
Measure: Number; unit: count of medication discrepancies
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone
Number analyzed (Participants) | 52 | 72
count of medication discrepancies | 63 | 81

4. Secondary Outcome: Care Transitions Measure Score
Description: A measure of condition self-knowledge and transitional care quality from the patient's perspective is ascertained by patient or caregiver interview 30 days after non-VA hospital discharge. The investigators will use an adapted 3-item version which includes items such as: "After I left the hospital, I had all the information I needed to be able to take care of myself" with the response options strongly agree, agree, disagree, strongly disagree, and don't know. The investigators chose to use the 3-item rather than a 15-item version as the shorter instrument demonstrates excellent correlation with the longer version but with lower respondent burden. Unabbreviated scale title is "3-Item Care Transitions Measure" and minimum value is 1 and maximum value is 12. Higher scores mean a better transition/outcome.
Time Frame: 30 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone
Number analyzed (Participants) | 54 | 73
score on a scale | 3.0 [3.0 to 3.7] | 3.0 [3.0 to 3.7]

ADVERSE EVENTS:
Time Frame: 90 days
Description: Participants were assessed for death regardless of whether or not they completed the study, whereas participants were assessed for Serious and Other (Not Including Serious) Adverse Events only if they completed the study. In addition, high-risk medication discrepancy was not assessed in the Usual Care group.
Arm/Group | HIE Notification Plus Care Coordination | HIE Notification Alone | Usual Care (No HIE Notification and No Care Coordination)
All-Cause Mortality (participants affected / at risk) | 20/268 | 31/337 | 26/191
Serious Adverse Events (participants affected / at risk) | 23/87 | 21/115 | 35/191
Other Adverse Events (participants affected / at risk) | 31/55 | 43/75 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIE Notification Plus Care Coordination (N=87) | HIE Notification Alone (N=115) | Usual Care (No HIE Notification and No Care Coordination) (N=191)
Hospital Readmission [Time frame 90 days] (Surgical and medical procedures) | 23 | 21 | 35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIE Notification Plus Care Coordination (N=55) | HIE Notification Alone (N=75) | Usual Care (No HIE Notification and No Care Coordination) (N=0)
Any high-risk medication discrepancy (Surgical and medical procedures) | 31 | 43 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT02689076/Prot_SAP_000.pdf